CLINICAL TRIAL: NCT04309786
Title: A Pilot Study of Somatization, Anxiety and Sleep Disorders in Pediatric Patients With Eosinophilic Esophagitis
Brief Title: Somatization, Anxiety, and Disordered Sleep in Pediatric Eosinophilic Esophagitis
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Principal Investigator, Seema Aceves, Professor, Pediatrics and Medicine, University of California, San Diego
Other Study IDs: 190374
Record Dates: First submitted 2019-06-27; First posted 2020-03-16 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Eosinophilic Esophagitis
Keywords: EoE
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eosinophilic esophagitis

DETAILED DESCRIPTION:
In order to decrease disease burden and the perception of disease burden, investigators need to understand the symptoms and severity of anxiety, disordered sleep, and somatization and how these parameters align with symptoms and quality of life in pediatric EoE. To assess the burden of these parameters in children with EoE, investigators will conduct a single center pilot study of 60 children with EoE using validated indexes for anxiety (state trait anxiety inventory for children), somatization (children's somatization inventory), sleep (pediatric sleep questionnaire), coping (Connor-Davidson Resilience Score) symptoms (PEESSv2.0), and quality of life (PedsQL-EoE).

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years old
* Ability to understand and complete the surveys and complete them in English
* Known diagnosis of EoE defined as > 15 eosinophils per high power field. Patient can have active or inactive disease at the time of entry

Exclusion Criteria:

* <8 or > 18 years old
* Inability to read the surveys in English
* Concurrent gastrointestinal diseases such as inflammatory bowel disease or Celiac disease.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children 8-18 years old seen in the Rady Children's EoE clinic population as part of routine care (n=60) patients
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Somatization score | Two weeks
  Our researchers will be using CSSI-Child Somatic Symptoms Inventory to measure the severity of bothersome somatic symptoms experienced in our EoE children and adolescents. Respondents are asked to rate the extent to which the child was bothered by each of the nonspecific somatic symptoms listed. Total scores are computed by summing the ratings for each item. Higher scores indicate greater somatic distress.
Sleep Quality score | Up to One month or in general
  Our researchers will be using PSQ-Pediatric Sleep Questionnaire to evaluate our EoE children's sleep disorder symptoms. This multi-page questionnaire consists of closed question-items and several open questions. The items are each answered yes = 1, no = 0, or don't know = missing. The number of symptom-items endorsed positively ("yes") is divided by the number of items answered positively or negatively; the denominator therefore excludes items with missing responses and items answered as don't know. The result is a number, a proportion that ranges from 0.0 to 1.0. Scores > 0.33 are considered positive and suggestive of high risk for a pediatric sleep-related breathing disorder
Anxiety score | At the moment and usually
  Our researchers will be using STAIC-State Trait Anxiety Questionnaire to evaluate. Our EoE children will be answering the questions in two different forms in which they report how they feel at a particular moment in time when they respond to the S-Anxiety scale (C-1), and how they generally feel when they respond to the T-Anxiety scale (C-2). Children respond to the STAIC by selecting one of the three alternative choices for each item which describes them best. In essence, each STAIC item is a 3-point rating scale for which values of 1, 2, or 3 are assigned for each of the three alternative choices. Thus, scores on both the STAIC S-Anxiety and T-Anxiety sub-scales can range from a minimum of 20 to a maximum score of 60. Higher scores mean higher anxiety.
Resilience score | One Month
  Connor-Davidson Resilience Scale (CD-RISC), We will be using this uni-dimensional self-reported scale to measure resilience in our EoE patients. Subjects will be responding to 10 items on a 5-point likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). Each item has a minimum score of 0 and a maximum score of 4. The total scores for this questionnaire range from a minimum of 0 to maximum of 40. The total scores are calculated by summing all 10 items. A higher score indicates higher resilience. None of the items are reverse scored.
Symptoms score | One month
  Our researchers will be using the Pediatric Eosinophilic Esophagitis Symptom Score (PEESSv2.0) to measure the severity and frequency of patient-relevant symptoms such as dysphagia, gastrointestinal reflux disease (GERD), nausea/vomiting, and pain. The PEESsv2.0 is a content-validated metric that seeks to capture EoE-specific symptoms directly from children with EoE (8-18 years of age) and from their parents (2-18 years of age). From parent/participant answers, four domains are evaluated: dysphagia, gastroesophageal reflux disease (GERD), nausea/vomiting and pain. The range for these PEESS® v2.0 scores are 0 to 100, with a higher score being indicative of more frequent and/or severe symptoms for total score, and the dysphagia, GERD, nausea/vomiting and pain domains.
Quality of Life score | One Month
  Our researchers will be using PedsQL-EoE questionnaire to measure different dimensions of EoE such as symptoms, treatment, worry, communication, food and eating, and food feelings. Children and parents answer 33 items comprising 7 dimensions mentioned above. Items are 5-point Likert scale from 0(never) to 4 (Almost Always). Scores are transformed on a scale from 0 to 100. Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. The mean score = Sum of the items over the number of items answered. Symptoms Total Scale Score can be obtained by Sum of the items over the number of items answered in the Symptoms I and Symptoms II Scales. The total Score can be obtained by sum of all the items over the number of items answered on all the Scales except Feeding Tube Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No